CLINICAL TRIAL: NCT06786351
Title: Impact of Right Atrial Occlusion on TEVAR Outcomes: A Prospective Cohort Study
Brief Title: Impact of Right Atrial Occlusion on TEVAR Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Claire Allen, Clinical Lecturer, University of Calgary
Other Study IDs: REB24-1367
Record Dates: First submitted 2025-01-07; First posted 2025-01-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Thoracic Aortic Aneurysm; Thoracic Aortic Dissection; Thoracic Aorta Abnormality
Keywords: right atrial balloon occlusion; thoracic endovascular aortic repair; stent graft repair; reduction of elimination of aortic impulse
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Dissection, Thoracic Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Right atrial balloon occlusion: Thoracic endovascular aortic repair with right atrial balloon occlusion for reduction or elimination of aortic impulse
  Interventions: Procedure: Right atrial balloon occlusion
- Non right atrial balloon occlusion: Thoracic endovascular aortic repair not using right atrial balloon occlusion for reduction or elimination of aortic impulse
  Interventions: Procedure: Non right atrial balloon occlusion

INTERVENTIONS:
Procedure: Right atrial balloon occlusion — Thoracic endovascular aortic repair with right atrial balloon occlusion for reduction or elimination of aortic impulse and stent graft deployment in landing zones 0-3
  Groups: Right atrial balloon occlusion
Procedure: Non right atrial balloon occlusion — Thoracic endovascular aortic repair not using right atrial balloon occlusion for reduction or elimination of aortic impulse and stent graft deployment in landing zones 0-3
  Groups: Non right atrial balloon occlusion

SUMMARY:
Though the application of thoracic endovascular aortic repair (TEVAR) for treatment of aortic pathology is expanding, there remains a gap in the literature examining how intraoperative "reduction or elimination of aortic impulse" (REAI) techniques, in particular the use of right atrial occlusion, may impact patient important clinical outcomes. This study aims to provide prospective data from a large cohort of TEVAR patients to explore clinical outcomes following TEVAR procedures and, specifically, whether right atrial occlusion has significant impact on clinical outcomes, as compared to other REAI techniques. The results from this study may inform future perioperative TEVAR practices and improve TEVAR patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* thoracic endovascular aortic repair
* right atrial balloon occlusion for reduction or elimination of aortic impulse
* endograft deployment in landing zones 0-3

Exclusion Criteria:

* age 18 years or younger
* non-thoracic endovascular aortic repair
* reduction or elimination of aortic impulse using technique other than right atrial balloon occlusion
* endograft deployment in landing zones 4 and beyond

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing emergency or elective thoracic endovascular aortic repair at the Peter Lougheed Centre, Calgary, Alberta
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Endoleak occurrence up to hospital discharge | end of surgery to hospital discharge up to 10 days)
  Endoleak occurrence prior to hospital discharge
Endoleak occurrence to one-year post-surgery | end of surgery to one-year post-surgery
  Endoleak occurrence within one-year of surgery

SECONDARY OUTCOMES:
Perioperative mortality to 30 days post-surgery | post-surgery to 30 days post-surgery
  30-day perioperative mortality
All-cause mortality to one-year post-surgery | post-surgery to one-year post-surgery
  One-year all-cause mortality
Complications: massive hemorrhage | within 30 days post-surgery and at 1 year
  Occurrence of massive hemorrhage
Complications: cerebrovascular | within 30 days post-surgery and at 1 year
  Occurrence of cerebrovascular accident/transient ischemic attack
Complications: spinal cord ischemia | within 30 days post-surgery and at 1 year
  Occurrence of spinal cord ischemia
Complications: iliofemoral access | within 30 days post-surgery and at 1 year
  Occurrence of iliofemoral access complications (bleeding/infection/thrombosis)
Complications: retrograde dissection | within 30 days post-surgery and at 1 year
  Occurrence of retrograde dissection
Complications: prolonged ventilation | within 30 days post-surgery and at 1 year
  Occurrence of prolonged ventilation for more than 24 hours
Complications: acute kidney injury | within 30 days post-surgery and at 1 year
  Occurrence of acute kidney injury
Complications: acute kidney injury with renal replacement therapy | within 30 days post-surgery and at 1 year
  Occurrence of acute kidney injury requiring renal replacement therapy
Complications: cardiovascular events | within 30 days post-surgery and at 1 year
  Occurrence of cardiovascular events (myocardial injury after non-cardiac surgery/cardiac arrest/myocardial infarction)